CLINICAL TRIAL: NCT00071565
Title: Familial Intracranial Aneurysm Study II
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Joseph Broderick, Joseph P. Broderick, University of Cincinnati
Other Study IDs: R01NS039512 (NIH); R01NS039512-06A1 (NIH)
Record Dates: First submitted 2003-10-28; First posted 2003-10-29 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Intracranial Aneurysm; Subarachnoid Hemorrhage
Keywords: familial intracranial aneurysm; intracranial aneurysm; brain aneurysm; aneurysm; subarachnoid hemorrhage; stroke
MeSH Terms: conditions — Intracranial Aneurysm; Subarachnoid Hemorrhage; Aneurysm; Stroke

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: 475 families with multiple affected family members (phase I) 200 families with multiple affected family members (phase II) 1800 subjects with sporadic intracranial aneurysms

SUMMARY:
The purposes of this study are to identify possible genes that may increase the risk of aneurysm development in the brain, and to determine the effect of environmental factors such as cigarette smoking and high blood pressure on the expression of these genes.

DETAILED DESCRIPTION:
Intracranial aneurysms are "blisters" which form within the arteries at the base of the brain. A rupture of an aneurysm may lead to subarachnoid hemorrhage (SAH). The mortality rates of patients suffering from a SAH is 40 to 44 percent , with many survivors enduring major disability. Most of the deaths from SAH are due to rapid and massive brain injury from the initial bleeding, which is not correctable by medical and surgical intervention. Thus, prevention of aneurysm formation is of paramount importance.

Scientific evidence suggests that a genetic component plays an important role in the development of intracranial aneurysms, however the specific genes have not been identified. The Familial Intracranial Aneurysm Study is a collaborative research effort of neurologists and neurosurgeons throughout the United States, Canada, Australia and New Zealand to identify possible genes that may increase the risk of stroke, and particularly, the development of aneurysms in the blood vessels of the brain. This study will involve 475 families with multiple affected family members, and will also determine the effect of environmental factors such as cigarette smoking and high blood pressure on the expression of the genes.A group of physicians from throughout North America, Australia and New Zealand have formed a collaborative effect to identify genes that may be important in the development of aneurysms in the blood vessels of the brain. This study of affected individuals and families, known as the Familial Intracranial Aneurysm (FIA) study, is sponsored by the National Institutes of Health and has involved over 475 families.

FIA II will involve an additional 200 families plus 1800 subjects with an Intracranial Aneurysm but no family history. These families and individuals will be used to replicate the findings of FIA I. FIA II will take place in North America only.

To be eligible to participate in this study, families must have two or more affected pairs of siblings (brothers/sisters) or 3 or more family members affected with intracranial aneurysms. Subjects can participate if they do not have an eligible family history, but do have a confirmed intracranial aneurysm.

Participants will be asked to complete a family history questionnaire (if they have a family history) and a medical history questionnaire. They will also have their blood pressure measured and will give a small sample of blood. In addition, medical records will be requested to confirm the diagnosis of intracranial aneurysms. There will be no monetary compensation for participation.

The identification of susceptibility genes, along with a better understanding of environmental interactions such as cigarette smoking, may result in preventing the development of intracranial aneurysms and/or intracranial aneurysm ruptures in people who are at risk for this condition.

ELIGIBILITY:
Inclusion:

* To be eligible to participate in this study, families must have two or more affected pairs of siblings (brothers/sisters) or 3 or more family members affected with intracerebral aneurysms.

Sporadic aneurysm subjects must have a confirmed aneurysm.

Exclusion:

* A history of polycystic kidney disease, Marfan's Syndrome, Ehlers Danlos Syndrome, or fibromuscular dysplasia.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 475 families with multiple affected family members will be selected in this collaborative research effort of neurologists and neurosurgeons throughout the United States, Canada, Australia and New Zealand (completed during phase I) 200 Families with multiple affected family members located in North America, and an additional 1800 subjects with sporadic aneurysm without a qualifing family history.
Sampling Method: Non-Probability Sample
Enrollment: 5875 (Actual)
Dates: Start 2002-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P. Broderick, M.D., Principal Investigator — University of Cincinnati
Locations (16):
- United States (16):
  - University of Alabama, Birmingham, Alabama
  - University of California,, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Indianapolis Neurosurgical Group, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Columbia University,, New York, New York
  - University of Cincinnati, Department of Neurology, Cincinnati, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Sauerbeck L, Hornung R, Woo D, Moomaw CJ, Anderson C, Connolly ES, Rouleau GA, Brown RD Jr, Broderick JP; FIA Study Investigators. Mortality and causes of death in the Familial Intracranial Aneurysm study. Int J Stroke. 2013 Dec;8(8):696-700. doi: 10.1111/j.1747-4949.2012.00857.x. Epub 2012 Aug 29. PMID 22928607